CLINICAL TRIAL: NCT00910000
Title: Phase Ib/II Study of Combination of Vorinostat, Carboplatin and Gemcitabine + Vorinostat Maintenance in Women With Recurrent, Platinum-Sensitive Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer
Brief Title: Vorinostat, Carboplatin and Gemcitabine in Women With Recurrent, Platinum-Sensitive Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to unacceptable toxicity
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Medical Director, Gynecologic Oncology, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-026
Record Dates: First submitted 2009-05-26; First posted 2009-05-29 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: carboplatin; gemcitabine; vorinostat
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Vorinostat; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose Level 1A (Experimental): Vorinostat: 200 mg taken orally once a day for the first two weeks of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 1 of every three week cycle
  Gemcitabine: 100 mg/m2, given intravenously on day 1 and day 8 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine
- Dose Level 2A (Experimental): Vorinostat: 300mg, taken orally once a day for the first two weeks of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 1 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 1 and day 8 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine
- Dose Level 1B (Experimental): Vorinostat: 200mg, taken orally twice a day for days 1-3 and days 8-10 of every three week cycle
  Carboplatin: AUC 4, given intravenously on day 1 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 1 and day 8 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine
- Dose Level 1C (Experimental): Vorinostat: 200mg, taken orally twice a day for days 1, 2, 8 and 9 of every three week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine
- Dose Level 1D (Experimental): Vorinostat: 300mg, taken orally once a day for days 1 and 2 of every three week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine
- Dose Level 2D (Experimental): Vorinostat: 400mg, taken orally once a day for days 1 and 2 of every three week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Vorinostat; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Vorinostat
  Other Names: Zolinza
Drug: Carboplatin
  Other Names: paraplatin
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
This trial is a Phase Ib/II study of carboplatin/gemcitabine/vorinostat for the treatment of platinum sensitive recurrent ovarian cancer. The carboplatin and gemcitabine combination is an FDA approved regimen for platinum-sensitive recurrent ovarian cancer. Vorinostat is a type of drug called a histone deacetylase inhibitor (HDAC inhibitor). HDAC inhibitors interact with chromosomes in the cancer cell and cause cancer cells to stop growing. Vorinostat has shown a decrease in the amount of ovarian cancer cells growing in the laboratory and also may enhance the anti-cancer effects of carboplatin.The purpose of the Phase Ib study is to determine the highest dose of the drug vorinostat that can be given safely in combination with carboplatin and gemcitabine. Not everyone who participates in this research study will receive the same dose of the study drug, vorinostat, but carboplatin and gemcitabine doses are held constant. Vorinostat doses depend on previous enrollment and tolerability. The expansion Phase II study uses the vorinostat dose found in the Phase Ib study in combination with carboplatin/gemcitabine and as a single agent maintenance therapy to better understand toxicity and efficacy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Phase Ib: Determine the maximally tolerated dose (MTD) of vorinostat when used in combination with standard (fixed) doses of carboplatin/gemcitabine during a 21 day cycle in patients with recurrent platinum-sensitive ovarian cancer

Phase II: Estimate the median progression-free survival (PFS) of patients treated with carboplatin/gemcitabine/vorinostat and vorinostat maintenance

Secondary

* Estimate the response rate of carboplatin/gemcitabine/vorinostat
* Assess the toxicities of carboplatin/gemcitabine/vorinostat
* Assess the toxicities of maintenance vorinostat
* Measure overall survival (OS) and progression-free survival (PFS)

STATISTICAL DESIGN:

The Phase Ib study was originally design to follow a standard 3+3 dose escalation design and evaluate 4 vorinostat dose levels.The DLT observation period was the 21-day cycle 1 length. Note: Ultimately 6 dose levels were evaluated as the protocol was amended to add dose levels, de-escalating cumulative vorinostat dose per cycle when 2 of 3 participants in dose level cohorts 2A, 1B and 1C experienced DLTs.

In the Phase II study, a median PFS of 13 months would be worthy of further study, representing a 66% improvement compared with the historical median of 8.6 months observed with carboplatin/gemcitabine. With 36 evaluable patients, there is 80% power to reject the null hypothesis in favor of the alternative at a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent epithelial ovarian cancer, fallopian tube cancer, or peritoneal cancer
* Must have received a platinum-based chemotherapy regimen at initial diagnosis
* Patients with primary platinum-sensitive (defined as a cancer initially platinum-sensitive followed by a progression-free interval from first exposure to platinum of 6 months or greater) recurrent ovarian, tubal or peritoneal cancer
* Must have an elevated CA125 (twice the ULN) within 2 weeks of enrolling on study (2 pretreatment measurements that are twice the upper limits of institutional normal and are drawn at least 1 day but not more than 14 days apart). At least one of the samples should be checked within one week of starting treatment. Measurable cancer via RECIST criteria via CT or MRI scan is not required but if clinically indicated will be monitored.
* For patients who do not have an elevated CA125 (twice the ULN), participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20mm or greater with conventional techniques or as 10mm or greater with spiral CT scan.
* 18 years of age or older
* Life expectancy of greater than 16 weeks
* ECOG Performance Status 0, 1, or 2
* Participants must have normal organ and marrow function as outlined in the protocol
* Patients could have received up to 1 prior non-platinum chemotherapy regimen in the recurrent setting (anti-angiogenic agents and other phase II non-hormonal therapies used to treat recurrent cancer count as a prior non-platinum therapy) but only one prior platinum (used to treat initial diagnosis). Patients may received up to 2 prior hormonal therapies.
* Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation
* Must be able and willing to take oral medications
* No clinical nor radiographic evidence of an existing or impending bowel obstruction
* Should be at least 2 weeks from any surgical procedure, with the exception of minor surgery, such as port placement
* Patients who have known carboplatin hypersensitivity reaction can receive carboplatin if they are followed by an allergist, follow a published hypersensitivity desensitization protocol when receiving carboplatin, and agree to receive carboplatin under these circumstances
* Patients taking valproic acid for epilepsy may enroll if they discontinue valproic acid 30 days prior to enrolling for washout
* Patients must have a normal QTc interval and no history of QTc prolongation on EKG

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* May not be receiving any other investigational agent
* Participants with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, pulmonary disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Individuals with a history of different malignancy are ineligible except for the following circumstances: disease-free for at least 5 years and are deemed by the investigator to be a low risk for recurrence of that malignancy; cervical cancer in situ, concurrent stage IA and grade I endometrial cancer, and basal cell or squamous cell carcinoma of the skin
* Patients taking valproic acid unless valproic acid is stopped at least 30 days prior to enrollment
* Receipt in the past of any other HDAC inhibitor for treatment of any malignancy
* Receipt of radiation therapy to >25% of bone marrow-bearing areas
* Patients who have gastrointestinal disorders likely to interfere with absorption of vorinostat
* Known active HIV or hepatitis viral infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A. Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matulonis U, Berlin S, Lee H, Whalen C, Obermayer E, Penson R, Liu J, Campos S, Krasner C, Horowitz N. Phase I study of combination of vorinostat, carboplatin, and gemcitabine in women with recurrent, platinum-sensitive epithelial ovarian, fallopian tube, or peritoneal cancer. Cancer Chemother Pharmacol. 2015 Aug;76(2):417-23. doi: 10.1007/s00280-015-2813-9. Epub 2015 Jun 29. PMID 26119093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants were enrolled and treated between July 2009 and January 2013. One patient excluded from all analyses failed screening after consent because of elevated liver function tests and did not receive treatment.
Period: Overall Study
Arm/Group | Dose Level 1A | Dose Level 2A | Dose Level 1B | Dose Level 1C | Dose Level 1D | Dose Level 2D
Started | 3 | 3 | 3 | 2 | 3 | 1
Completed | 3 | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 3 | 3 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 3 | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1B: Vorinostat: 200mg, taken orally twice a day for days 1-3 and days 8-10 of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 1 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 1 and day 8 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
- Dose Level 1C: Vorinostat: 200mg, taken orally twice a day for days 1, 2, 8 and 9 of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
- Dose Level 1D: Vorinostat: 300mg, taken orally once a day for days 1 and 2 of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
- Dose Level 2D: Vorinostat: 400mg, taken orally once a day for days 1 and 2 of each three-week cycle
  Carboplatin: AUC 4, given intravenously on day 2 of every three week cycle
  Gemcitabine: 1000 mg/m2, given intravenously on day 2 and day 9 of every three week cycle
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1A | Dose Level 2A | Dose Level 1B | Dose Level 1C | Dose Level 1D | Dose Level 2D | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 1 | 15
Age, Customized [Mean (Full Range); unit: years]
  Age | 59 [51 to 68] | 63 [61 to 65] | 59 [54 to 66] | 54.5 [52 to 57] | 67 [58 to 75] | 63 [NA to NA] — There is only 1 patient in this cohort. | 60 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 3 | 1 | 15
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 2 | 3 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Vorinostat Maximum Tolerated Dose (MTD) [Phase Ib]
Description: The Vorinostat MTD is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached.
Time Frame: The DLT observation period in determining the MTD was the 21-day cycle 1 length.
Population: Per protocol, MTD evaluable participants received day 1 of treatment, were not taken off study during cycle 1 due to disease progression, showed proof via pill diary that all doses of vorinostat were taken or attempted to be taken and were compliant with study procedures. The final MTD dataset was comprised of all enrolled and treated participants.
Measure: Number; unit: mg/day
Groups:
- All Phase Ib Participants: All Phase Ib participants received Vorinostat according to the established dose escalation schedule during a 3-week cycle in combination with IV carboplatin AUC 4 (day 2) and IV gemcitabine 1000 mg/m2 (days 2 and 9).
  Participants received up to 8 cycles of therapy without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
Arm/Group | All Phase Ib Participants
Number analyzed (Participants) | 15
mg/day | NA — Protocol was amended to add reduced V. total dose when 2 of 3 participants in DL 2A, 1B & 1C experienced DLTs. MTD was not reached w/ the study term early due to safety concerns when the first patient in the dose level cohort 2D experienced a DLT.

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase Ib]
Description: Dose-limiting toxicity was based on the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) and defined as any of the following:
  1. Any CTCAE grade 3 or 4 non-hematologic event except manageable gastrointestinal toxicity and fatigue.
  2. Any of the following hematologic events (excluding neutropenia lasting < 5 days):
     i) febrile neutropenia defined as grade 3-4 neutropenia with fever ≥ 38.5°C and/or infection.
     ii) any grade 4 neutropenia lasting 5 days or more. iii) grade 4 thrombocytopenia (plt count < 25x 109/L) iv) failure of ANC to recover to ≥ 1000/μL or platelets to recover to ≥ 50,000/μL within 14 days of therapy v) grade 4 anemia
  3. Any clinically significant abnormal laboratory value that results in dose delay of >14 days.
  4. <75% of vorinostat dosing taken by the patient during the first cycle due to any toxicity.
Time Frame: The DLT observation period in determining the MTD was the 21-day cycle 1 length.
Population: Per protocol, DLT evaluable participants received day 1 of treatment, were not taken off study during cycle 1 due to disease progression, showed proof via pill diary that all doses of vorinostat were taken or attempted to be taken and were compliant with study procedures. The final DLT dataset was comprised of all enrolled and treated participants.
Measure: Number; unit: participants with DLT
Arm/Group | Dose Level 1A | Dose Level 2A | Dose Level 1B | Dose Level 1C | Dose Level 1D | Dose Level 2D
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 1
participants with DLT | 0 | 2 | 2 | 2 | 0 | 1

3. Secondary Outcome: Response
Description: Response was based on RECIST 1.0 criteria. Per RECIST 1.0 for target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD from the smallest LD recorded on treatment. Stable disease (SD) is neither sufficient increase to qualify as PD nor sufficient shrinkage to qualify for PR. For CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed 4 weeks +/- 2 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Participants who received therapy but did not have their disease re-evaluated were considered unevaluable.
Time Frame: Disease was assessed radiographically (CT or MRI scan) every 2 cycles on treatment; Phase Ib participants received up to 8 cycles of treatment. The median number of cycles started was 2 (range 1-8).
Measure: Number; unit: participants
Arm/Group | Dose Level 1A | Dose Level 2A | Dose Level 1B | Dose Level 1C | Dose Level 1D | Dose Level 2D
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 1
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 3 | 0 | 0 | 1 | 2 | 0
  Stable Disease | 0 | 1 | 0 | 0 | 0 | 0
  Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0
  Unevaluable | 0 | 2 | 3 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every cycle on treatment. Phase Ib participants received up to 8 cycles of treatment. The median number of cycles started was 2 (range 1-8).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | All Phase Ib Participants
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Phase Ib Participants (N=15)
Fatigue (General disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 9
Platelets (Blood and lymphatic system disorders) | 8
Leukocyte (Blood and lymphatic system disorders) | 2
Allergic Reactions (Immune system disorders) | 1
Pulmonary Embolism (Vascular disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Phase Ib Participants (N=15)
Neutropenia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 12
Nausea (Gastrointestinal disorders) | 13
Platelets (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Hypomagnesemia (Investigations) | 5
Leukocyte (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Alopecia (General disorders) | 3
Allergic Reactions (Immune system disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Neuropathy (Nervous system disorders) | 2
Phlebitis (General disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated early for toxicities and the emergence of better tolerated and more promising biologic agents added to platinum-based chemotherapy and/or use as maintenance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less